CLINICAL TRIAL: NCT06551623
Title: A Single Center, Open Label, Phase 1 Study in Healthy Participants to Investigate the Drug-Drug Interactions Between TNP-2198 and Midazolam, Clarithromycin
Brief Title: Drug-Drug Interactions Between TNP-2198 and Midazolam, Clarithromycin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TenNor Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TNP-2198-10
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Midazolam; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Midazolam cohort (Experimental): Midazolam Oral Solution will be given orally once daily within 0.5 hours after breakfast on Day 1 and Day 10.
  TNP-2198 Capsules will be given orally twice daily within 0.5 hours after breakfast and dinner from Day 3 to Day 11.
  Interventions: Drug: Midazolam; Drug: TNP-2198
- Clarithromycin cohort (Experimental): Clarithromycin tablets will be given orally within 0.5 hours after breakfast and dinner from Day 16 to Day 25.
  TNP-2198 Capsules will be given orally twice daily within 0.5 hours after breakfast and dinner from Day 1 to Day 7 and from Day16 to Day 22, and once daily within 0.5 hours after breakfast on Day 8 and Day 23.
  Interventions: Drug: Clarithromycin; Drug: TNP-2198

INTERVENTIONS:
Drug: Midazolam — Midazolam Oral Solution 2 mg
  Arms: Midazolam cohort
Drug: Clarithromycin — Clarithromycin tablets 0.5 g
  Arms: Clarithromycin cohort
Drug: TNP-2198 — TNP-2198 Capsules 400 mg

SUMMARY:
This is a single center, open label, drug-drug interaction, Phase 1 study of TNP-2198 in approximately 32 healthy participants, includes 2 cohorts (16 participants per cohort): Midazolam cohort and Clarithromycin cohort. Midazolam cohort will evaluate the effect of multiple oral doses of TNP-2198 capsules on the pharmacokinetics (PK) parameters of a single oral dose of midazolam, a cytochrome P-450 (CYP) 3A sensitive substrate, in healthy participants; Clarithromycin cohort will evaluate the effect of multiple oral doses of clarithromycin tablets, a strong CYP3A and P-gp inhibitor, on the PK parameters of multiple oral doses of TNP-2198 in healthy participants.

DETAILED DESCRIPTION:
Midazolam cohort: Midazolam oral solution will be administered orally at a dose of 2 mg once a day within 0.5 hours after breakfast on Day 1, and administered following TNP-2198 capsules within 0.5 hours after breakfast on Day 10. TNP 2198 capsules will be administered orally at a dose of 400 mg twice a day, within 0.5 hours after breakfast and dinner, from Day 3 to Day 11. PK blood sampling and safety tests were performed at specified time points.

Clarithromycin cohort: TNP-2198 capsules will be administered orally at a dose of 400 mg twice a day, within 0.5 hours after breakfast and dinner, from Day 1 to Day 7, and within 0.5 hours after breakfast on Day 8. Clarithromycin tablets will be administered at a dose of 0.5 g twice a day, within 0.5 hours after breakfast and dinner, from Day 16 to Day 25. TNP-2198 capsules will be administered within 0.5 hours after breakfast and dinner, followed by clarithromycin tablets, from Day 16 to Day 22. TNP-2198 capsules will be administrated within 0.5 hours after breakfast, followed by clarithromycin tablets on Day 23. PK blood sample collection and safety tests were performed at specified time points.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide written Informed consent forms (ICF) and fully understand the study procedures and potential AEs.
* Be able to comply with all protocol requirements.
* Willing to voluntarily take effective contraceptive measures from signing the ICF to 3 months after the last dose of investigational product, and male subjects must refrain from sperm donation during this period.
* Male or female, 18 to 55 years of age, inclusive.
* Have a body mass index (BMI) 18 to 28 kg/m2, inclusive, and body weight ≥ 50 kg for male or ≥ 45 kg for female.
* The results of physical examination and vital signs are normal or abnormal but without clinical significance.

Exclusion Criteria:

* Have a history of allergy to the investigational products (TNP-2198, midazolam [Midazolam cohort] or clarithromycin [Clarithromycin cohort]), and/or allergic constitution (such as allergic to multiple drugs, food or pollen, or prone to allergic reactions without knowing the causes of allergy).
* Have abnormal laboratory tests with clinical significance, or have dysphagia, or have diseases that can affect drug absorption or excretion within 6 months before screening, or other clinical findings within 12 months before screening indicating clinically significant diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases.
* Have an abnormal result of ECG with clinical significance at screening/baseline.
* Have a positive test result for Hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), AIDS antibody or Treponema pallidum antibody at screening/baseline.
* Female participants have a positive result for pregnancy test at screening or admission or are lactating.
* Have a positive result for orthostatic hypotension at screening, or have a history of orthostatic hypotension, when screening for Midazolam cohort.
* Have used CYP3A inducers or inhibitors (such as clarithromycin, erythromycin, verapamil, diltiazem, ketoconazole, itraconazole, ritonavir, etc.), P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP) inhibitors or inducers (such as itraconazole, ketoconazole or dronedarone, etc.) within 30 days before screening.
* Participants who must take prescription or non-prescription drugs (including vitamins and dietary or herbal supplements, etc.) within 7 days or 5 half-lives (whichever is longer) before the administration of investigational products or throughout the study, unless the investigator considers that the drug will not interfere with the study. Any exceptions will be discussed with the sponsor case-by-case and the reasons will be documented.
* Participants enrolled in other clinical trials, or received other investigational products, or used medical devices within 3 months before the administration of investigational products in this study, or 5 half-lives of other investigational products, or twice the duration of biological effect of other investigational products (whichever is longer).
* Smoke more than 5 cigarettes or equivalent cigarettes per day on average within 3 months prior to the first dose, or unable to stop smoking during the study.
* Have alcohol abuse within 6 months before screening, that is, drink more than 14 units of alcohol per week on average (1 unit = 285 mL of beer, or 45 mL of 40% liquor, or 100 mL of wine), or cannot stop drinking any alcohol-containing products during the study, or drinking or taking any alcohol-containing products within 48 hours before the first dose, or alcohol breath test result is positive at screening/baseline.
* Have a history of drug abuse within 6 months prior to screening or have positive results for drug screening tests at baseline.
* Have received live or attenuated vaccines within 1 month before screening, or plan to receive live or attenuated vaccines during the study.
* Have a blood donation more than 400 mL within 3 months before the first dose of investigational products or have received a blood transfusion within 1 month before screening.
* Have special food (such as chocolate, dragon fruit, mango, grapefruit, any diet containing caffeine or xanthine) or be involved in strenuous exercise within 48 hours before the first dose of investigational product.
* Have an acute disease or concomitant medication from the screening period to before taking the investigational products.
* Have acute angle-closure glaucoma or open angle glaucoma without effective treatment at screening for Midazolam cohort.
* Have a history of congenital or acquired QT prolongation, or ventricular arrhythmia history at screening for Clarithromycin cohort.
* The investigator considers that the participant is unable to comply with all study procedures, or has other conditions that are not suitable for participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Midazolam cohort: PK parameters of midazolam-Area under the plasma concentration versus time curve (AUC0-t) | Within 1 hour prior to midazolam dosing and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours following midazolam dosing on Day 1 and Day 10, respectively.
  Area under the plasma concentration versus time curve from time 0 to the last quantifiable concentration (AUC0-t)
Midazolam cohort: PK parameters of midazolam-Area under the plasma concentration versus time curve (AUC0-∞) | Within 1 hour prior to midazolam dosing and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours following midazolam dosing on Day 1 and Day 10, respectively.
  Area under the plasma concentration versus time curve from time 0 extrapolated to infinity (AUC0-∞)
Midazolam cohort: PK parameters of midazolam-Maximum observed plasma concentration (Cmax) | Within 1 hour prior to midazolam dosing and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours following midazolam dosing on Day 1 and Day 10, respectively.
  Maximum observed plasma concentration (Cmax)
Clarithromycin cohort: PK parameters of TNP-2198-Area under the plasma concentration versus time curve(AUC0-t) | Within 1 hour prior to TNP-2198 dosing and at 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, and 72 hours following TNP-2198 dosing on Day 8 and Day 23, respectively.
  Area under the plasma concentration versus time curve from time 0 to the last quantifiable concentration
Clarithromycin cohort: PK parameters of TNP-2198-Area under the plasma concentration versus time curve from time 0 extrapolated to infinity (AUC0-∞) | Within 1 hour prior to TNP-2198 dosing and at 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, and 72 hours following TNP-2198 dosing on Day 8 and Day 23, respectively.
  Area under the plasma concentration versus time curve from time 0 extrapolated to infinity
Clarithromycin cohort: PK parameters of TNP-2198-Maximum observed plasma concentration (Cmax) | Within 1 hour prior to TNP-2198 dosing and at 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, and 72 hours following TNP-2198 dosing on Day 8 and Day 23, respectively.
  Cmax

SECONDARY OUTCOMES:
Midazolam cohort: Percentage of Participants With Adverse Events (AEs) | Day 1 to Day 12
  An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events
Clarithromycin cohort:Percentage of Participants With Adverse Events (AEs) | Day 1 to Day 26
  An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events
Midazolam cohort: PK parameters of midazolam Time to Maximum Plasma Concentration (Tmax) | Within 1 hour prior to midazolam dosing and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours following midazolam dosing on Day 1 and Day 10, respectively.
  Time to Maximum Plasma Concentration (Tmax)
Midazolam cohort: PK parameters of midazolam Terminal Elimination Half-life (T1/2) | Within 1 hour prior to midazolam dosing and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours following midazolam dosing on Day 1 and Day 10, respectively.
  Terminal Elimination Half-life (T1/2)
Clarithromycin cohort: PK parameters of TNP-2198 Time to Maximum Plasma Concentration (Tmax) | Within 1 hour prior to TNP-2198 dosing and at 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, and 72 hours following TNP-2198 dosing on Day 8 and Day 23, respectively.
  Time to Maximum Plasma Concentration (Tmax)
Clarithromycin cohort: PK parameters of TNP-2198 Terminal Elimination Half-life (T1/2) | Within 1 hour prior to TNP-2198 dosing and at 1, 2, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, and 72 hours following TNP-2198 dosing on Day 8 and Day 23, respectively.
  Terminal Elimination Half-life (T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojiao Li, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jinlin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No